CLINICAL TRIAL: NCT03087721
Title: Efficacy of High-intensity Interval, Low-volume Training Compared to Continuous Aerobic Exercise on Insulin Resistance, Skeletal Muscle Composition and Endocrine Function in Adults With Metabolic Syndrome: a Randomized Controlled Clinical Trial (Intraining-MET)
Brief Title: High-intensity Interval, Low Volume Training in Metabolic Syndrome
Acronym: Intraining-MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Principal Investigator, Jaime Gallo, MD, MSc, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54-2016
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Metabolic Syndrome; Insulin Resistance
Keywords: Metabolic Syndrome; Exercise Training; Interval Training; Skeletal Muscle; Risk Factors; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1x2 HIIT-LV, 3 times a week, 24 min (Experimental)
  Interventions: Behavioral: HIIT-LV
- CAE, moderate intensity, 3 times a week, 36 min (Active Comparator)
  Interventions: Behavioral: CAE

INTERVENTIONS:
Behavioral: HIIT-LV — Supervised endurance treadmill training as walking/running "uphill", 3 times/week during 12 weeks starting at 85-90% of previously determined maximum oxygen consumption (VO2 max). Warm-up 3 min at 30% of VO2 max, 3 min cool-down. Progression in intensity every 3erd week.
  Arms: 1x2 HIIT-LV, 3 times a week, 24 min
Behavioral: CAE — Supervised moderate intensity treadmill training, 3 times/week for 12 weeks starting at 70% of VO2 max. Warm-up 3 min at 30% of VO2 max, 3 min cool-down. Progression in intensity every 3erd week.
  Arms: CAE, moderate intensity, 3 times a week, 36 min

SUMMARY:
The primary objective of the study is to compare the efficacy of an intervention with high-intensity interval, low volume training (HIIT-LV) or continuous aerobic exercise (CAE) on insulin resistance, insulin sensitivity and percentage of pancreatic β-cell function in adults with metabolic syndrome (MS).

The secondary objective is to compare the efficacy of an intervention with HIIT-LV or CAE on glycosylated hemoglobin, mass and muscle fibre type composition of right thigh and plasma levels of musclin and apelin in adults with MS.

The investigators hypothesized that HIIT-LV is more effective in decreasing insulin resistance and glycosylated hemoglobin and plasma concentrations of musclin and increasing plasma concentrations of apelin, and both mass and muscle fibre type I percentage in thigh, than CAE.

DETAILED DESCRIPTION:
This study is a randomized, controlled, masked (single blind, outcomes assessor) clinical trial, with allocation by the minimization method, with two parallel groups and intention of superiority. It was designed to test the hypothesis that a 12-week program of HIIT-LV, yields larger beneficial effects on insulin resistance, skeletal muscle composition and endocrine function than CAE.

Although aerobic exercise increases cardio-respiratory capacity, modifies risk factors and decreases mortality risk, there is currently controversy and gaps in knowledge over the efficacy of more intense and low-volume physical activities on muscle metabolism in patients with metabolic disorders.

The primary outcome will be the insulin resistance, insulin sensitivity and percentage of pancreatic β-cell function. The secondary outcomes will be the glycosylated hemoglobin, mass and muscle fibre type composition of thigh and plasma levels of musclin and apelin. Assessments will be made before and after the 12-week program. Calculations based on previously results (difference mean 10% and SD 15%) suggest that a total number of 60 patients randomized 1:1 (30 in each group) to the two intervention groups is sufficient to detect larger beneficial effects with HIIT-LV with a p-value of 0.05 (two-sided test) and statistical power of 0.80 (primary endpoint is insulin sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome defined according to the International Diabetes Federation-criteria.
* Insulin resistance defined according to the HOMA greater than 2.25
* Sedentary lifestyle (less than 60 min of physical activity per week)

Exclusion Criteria:

* Vegetarian diet
* Vitamin D3 supplementation
* Oral contraceptives
* Musculoskeletal diseases or injuries
* Physical, sensory or cognitive impairment
* History of cardiovascular disease (coronary, cerebrovascular, peripheral arterial disease, uncontrolled cardiac arrhythmias).
* Pulmonary diseases
* Acute or chronic inflammatory conditions
* Cancer
* Human immunodeficiency virus infection
* Diabetes mellitus
* Hyperthyroidism
* Pregnancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 12-week
  Using HOMA model (units as percentages of a normal reference population)
Insulin resistance | 12-week
  Using HOMA model (arbitrary units)
Pancreatic β-cell function | 12-week
  Using HOMA model (units as percentages of a normal reference population)

SECONDARY OUTCOMES:
Glycosylated hemoglobin | 12-week
  Using blood tests (%)
Mass muscle of right thigh | 12-week
  Using dual energy x-ray absorptiometry (DEXA) (kg/m2)
Muscle fibre type composition of right thigh | 12-week
  Using carnosine quantification by hydrogen magnetic resonance spectroscopy (1H-MRS) (% fibre type I)
Musclin | 12-week
  Using plasma levels of musclin (pg/mL)
Apelin | 12-week
  Using plasma levels of apelin (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Calderón, MD, PhD, Principal Investigator — Professor; Daniel Aguirre, PhD, Study Director — Professor
Locations (1):
- IPS-Universitaria, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gallo-Villegas J, Restrepo D, Perez L, Castro-Valencia LA, Narvaez-Sanchez R, Osorio J, Aguirre-Acevedo DC, Calderon JC. Safety of High-Intensity, Low-Volume Interval Training or Continuous Aerobic Training in Adults With Metabolic Syndrome. J Patient Saf. 2022 Jun 1;18(4):295-301. doi: 10.1097/PTS.0000000000000922. Epub 2021 Sep 20. PMID 34870388
- [Derived] Aristizabal JC, Montoya E, Sanchez YL, Yepes-Calderon M, Narvaez-Sanchez R, Gallo-Villegas JA, Calderon JC. Effects of Low-Volume, High-Intensity Interval Training Compared with Continuous Training on Regional and Global Body Composition in Adults with Metabolic Syndrome: A post hoc Analysis of a Randomized Clinical Trial. Ann Nutr Metab. 2021;77(5):279-288. doi: 10.1159/000518909. Epub 2021 Oct 6. PMID 34763335
- [Derived] Gallo-Villegas J, Castro-Valencia LA, Perez L, Restrepo D, Guerrero O, Cardona S, Sanchez YL, Yepes-Calderon M, Valbuena LH, Pena M, Milan AF, Trillos-Almanza MC, Granados S, Aristizabal JC, Estrada-Castrillon M, Narvaez-Sanchez R, Osorio J, Aguirre-Acevedo DC, Calderon JC. Efficacy of high-intensity interval- or continuous aerobic-training on insulin resistance and muscle function in adults with metabolic syndrome: a clinical trial. Eur J Appl Physiol. 2022 Feb;122(2):331-344. doi: 10.1007/s00421-021-04835-w. Epub 2021 Oct 23. PMID 34687360
- [Derived] Gallo-Villegas J, Aristizabal JC, Estrada M, Valbuena LH, Narvaez-Sanchez R, Osorio J, Aguirre-Acevedo DC, Calderon JC. Efficacy of high-intensity, low-volume interval training compared to continuous aerobic training on insulin resistance, skeletal muscle structure and function in adults with metabolic syndrome: study protocol for a randomized controlled clinical trial (Intraining-MET). Trials. 2018 Feb 27;19(1):144. doi: 10.1186/s13063-018-2541-7. PMID 29482601